CLINICAL TRIAL: NCT01530295
Title: Biochemical Recurrence Rate of Radical Prostatectomy Combined With Neoadjuvant and Adjuvant in Patients With High Risk Locallized Prostate Cancer
Brief Title: Biochemical Recurrence Rate of Radical Prostatectomy Combined With Neoadjuvant and Adjuvant Chemotherapy in High Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanjong Ahn (Other)
Responsible Party: Sponsor-Investigator, Hanjong Ahn, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 2007-0326
Record Dates: First submitted 2011-06-22; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- contol (No Intervention): control group
  Interventions: Drug: DOCETAXEL
- chemotherapy (Other): neoadjuvant chemotherapy
  Interventions: Drug: DOCETAXEL

INTERVENTIONS:
Drug: DOCETAXEL — 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle. Number of Cycles: 3 times pre-op and 3 times after surgery
  Other Names: taxotere

SUMMARY:
Effect of Radical Prostatectomy Combined with Neoadjuvant and Adjuvant Chemotherapy in Patients with High Risk Prostate Cancer.

The purpose of this study is to evaluate whether neoajuvant and adjuvant docetaxel and prednisone are effective in the treatment of high risk localized prostate cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether neoajuvant and adjuvant docetaxel and prednisone are effective in the treatment of high risk localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer
* PSA > 20 OR
* Clinical Stage > T2C OR
* GS > 7

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
biochemical recurrence rate of Radical Prostatectomy Combined with Neoadjuvant and Adjuvant Chemotherapy in Patients with High Risk Prostate Cancer | 2 Years After RRP

CONTACTS AND LOCATIONS:
Overall Officials: hanjong Ahn, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Jungmin Lee, Seoul, Seoul, South Korea